CLINICAL TRIAL: NCT00677534
Title: Exploring the Role of Extrarenal 1-Alpha-Hydroxylase in Patients With End Stage Renal Disease
Brief Title: Role of Extrarenal 1-Alpha-Hydroxylase in Patients With End Stage Renal Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas (Other)
Responsible Party: Principal Investigator, Jason Stubbs, MD, Assistant Professor, University of Kansas
Organization: University of Kansas Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11225
Record Dates: First submitted 2008-05-12; First posted 2008-05-14 (Estimated); Results first posted 2014-03-21 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-04

CONDITIONS: End-Stage Renal Disease
Keywords: Endstage renal disease; Vitamin D; Monocyte function
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Cholecalciferol; Ergocalciferols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Cholecalciferol (Vitamin D)
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol — 50,000 Units PO Twice weekly for 8 weeks
  Other Names: Vitamin D, ergocalciferol

SUMMARY:
The goal of this study is to evaluate the role of nutritional Vitamin D deficiency as a potential contributor to the morbidity witnessed in patients with end-stage renal disease

DETAILED DESCRIPTION:
The goals of this study are to elucidate the function of extrarenal 1 alpha-hydroxylase activity in the setting of renal failure and to evaluate the role of nutritional vitamin D deficiency as a potential contributor to monocyte-associated inflammatory pathways in patients with end-stage renal disease (ESRD). This study will consist of patients on chronic maintenance hemodialysis three times per week who have been identified to have nutritional vitamin D deficiency. After consent for study enrollment, patients will undergo a 4 week washout period of all active vitamin D supplementation. After washout is complete, an blood sample will be obtained for baseline 25(OH)D levels and monocyte isolation for analysis by flow cytometry. Patients will then be started on cholecalciferol 50,000 IU twice weekly for 8 weeks. 25-vitamin D levels will be monitored midway through the treatment phase of the study and dosing adjusted as further described in detail within the protocol section. An additional blood sample will be drawn post-therapy for repeat 25(OH)D levels and monocyte isolation for flow cytometry analysis.

ELIGIBILITY:
Inclusion Criteria:

* End-stage renal disease undergoing maintenance hemodialysis at KUMC outpatient hemodialysis unit
* Dialysis vintage of at least 6 months duration
* Nutritional vitamin D deficiency, defined as 25(OH)D <25 ng/ml
* Age 21 to 88 years

Exclusion Criteria:

* Active infection
* Recent hospitalization for acute illness (within last 1 month)
* Refusal to study participation
* Poorly controlled secondary hyperparathyroidism (iPTH>500)
* History of chronic inflammatory disease process, such as inflammatory bowel, rheumatoid arthritis, lupus, etc.
* Cinacalcet therapy
* Previous allergy to ergocalciferol
* History of parathyroidectomy
* Current treatment with immunosuppressant medications
* Noncompliance with prescribed hemodialysis regimen (i.e. skipping treatments, ending sessions early)
* Functional renal transplant within the last five years

Ages: 21 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2008-05; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Stubbs, MD, Principal Investigator — University of Kansas Medical Center

REFERENCES:
- [Result] Stubbs JR, Idiculla A, Slusser J, Menard R, Quarles LD. Cholecalciferol supplementation alters calcitriol-responsive monocyte proteins and decreases inflammatory cytokines in ESRD. J Am Soc Nephrol. 2010 Feb;21(2):353-61. doi: 10.1681/ASN.2009040451. Epub 2009 Dec 10. PMID 20007751

RESULTS

PARTICIPANT FLOW:
Groups:
- Cholecalciferol 50,000 U: Vitamin D
Period: Washout (Weeks 1-4)
Arm/Group | Cholecalciferol 50,000 U
Started | 10
Completed | 7
Not Completed | 3
Not completed — did not qualify after signing consent | 1
Not completed — Withdrawal by Subject | 1
Not completed — Withdrawal by Subject | 1
Period: Cholecalciferol (Weeks 5-12)
Arm/Group | Cholecalciferol 50,000 U
Started | 7
Completed | 7
Not Completed | 0
Period: After Paricalcitol Restart (Weeks 13-14)
Arm/Group | Cholecalciferol 50,000 U
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: A total of 11 subjects were consented to the study. 1 subject was hospitalized before starting any procedures and did not complete any study procedures. 1 subject did not qualify for the study after consenting. Two subjects withdrew after consenting.
Arm/Group | Cholecalciferol 50,000 U
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 11
Monocyte Vitamin D receptor (VDR) expression [Mean (Standard Deviation); unit: MFI] | 572.7 (172.3)

OUTCOME MEASURES:

1. Primary Outcome: Change in Monocyte VDR Expression With Vitamin D Therapy
Description: Monocytes will be analyzed pre- and post-cholecalciferol by flow cytometry to measure changes in monocyte VDR expression. Unit of measure is represented by mean florescence intensity (MFI), which is a relative measure.
Time Frame: Change from End of Washout to Week 12
Population: Clinical pilot trial - proof of concept
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cholecalciferol 50,000 U
Number analyzed (Participants) | 7
units on a scale | 1899 (644.4)

ADVERSE EVENTS:
Arm/Group | Cholecalciferol 50,000 U
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

LIMITATIONS AND CAVEATS:
This was a pilot study using a small number of patients. Further studies are needed to validate these findings in larger groups of patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes